CLINICAL TRIAL: NCT00841152
Title: A National, Prospective, Randomized, Multicenter, Controlled Head-to-Head Comparison of Bioactive Glass and Beta-Tricalcium Phosphate as Bone Graft Substitute in Filling of Contained Bone Defects
Brief Title: Comparison of Bioactive Glass and Beta-Tricalcium Phosphate as Bone Graft Substitute
Acronym: BAGvsTCP
Status: Completed | Type: Observational
Sponsor: Turku University Hospital (Other Government)
Responsible Party: Sponsor
Other Study IDs: 139/180/2008
Record Dates: First submitted 2009-02-10; First posted 2009-02-11 (Estimated); Last update posted 2021-03-16 (Actual); Status verified 2021-03

CONDITIONS: Bone Neoplasm
Keywords: Bone tumors; Surgery; Bone graft substitutes; Bioactive glass; Bioceramics; Bone autograft; Bone allograft
MeSH Terms: conditions — Bone Neoplasms | interventions — Transplantation, Autologous; Transplantation, Homologous

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Hand lesions: Stratum I: comparison of three interventions (autograft, bioactive glass and beta-tricalcium phosphate)
  Interventions: Device: Bioactive glass; Device: Beta-tricalcium phosphate (ChronOs); Procedure: Autograft
- Long-bone lesions: Stratum II: comparison of three interventions (bioactive glass, beta-tricalcium phosphate, allograft)
  Interventions: Device: Bioactive glass; Device: Beta-tricalcium phosphate (ChronOs); Procedure: Allograft (frozen femoral head)

INTERVENTIONS:
Device: Bioactive glass — Surgical implantation
  Other Names: Bonalive (Vivoxid Ltd, Turku, Finland)
Device: Beta-tricalcium phosphate (ChronOs) — Surgical implantation
  Other Names: ChronOs (Synthes, Solothurn, Switzerland)
Procedure: Autograft — Surgical transplantation from iliac crest
  Groups: Hand lesions
Procedure: Allograft (frozen femoral head) — Surgical transplantation
  Groups: Long-bone lesions

SUMMARY:
This study is designed to perform a head-to-head comparison of two synthetic ceramic bone graft substitutes, bioactive glass (BAG) and beta-tricalcium phosphate (TCP), in filling of contained bone defects following surgical evacuation of benign bone tumor or tumor-like conditions. Based on the investigators' previous preclinical research and an ongoing single-center randomized clinical trial on bioactive glass filling, the investigators expect BAG filling to be more efficient compared to TCP in promotion of defect healing and functional recovery after surgery.

DETAILED DESCRIPTION:
This study is designed to perform a head-to-head comparison of two synthetic ceramic bone graft substitutes, bioactive glass (BAG) and beta-tricalcium phosphate (TCP), in filling of contained bone defects following surgical evacuation of benign bone tumor or tumor-like conditions. Small metacarpal and phalangeal enchondromas (Stratum I) and large long-bone lesions (Stratum II) will be evaluated separately. Aside with the head-to-head comparison of the two synthetic bone graft substitutes, autologous bone graft (Stratum I) and allogeneic bone graft (Stratum II) will be used as the standard of care controls.

ELIGIBILITY:
Inclusion Criteria:

* Patients with primary or recurrent benign bone tumor or tumor-like condition that requires operative treatment by means of tumor evacuation and defect filling
* Pathological fractures of patients in Stratum I are treated by means of conservative treatment for three months before tumor surgery

Exclusion Criteria:

* History of acute or chronic local infection
* History of malignancy (excluding carcinoma basocellular) within past 5 years
* A history of local radiotherapy
* A known metabolic skeletal disease (such as osteoporosis, Paget's disease or osteomalacia)
* Medication affecting bone turnover (oral bisphosphonates, PTH, sodium fluoride, strontium ranelate, calcitonin, testosterone, systemic cortico- or anabolic steroids)
* Any plans to use phenol or other chemical/thermal method of local tumor control
* Pregnancy
* Any other condition that in the judgment of the investigator, would prohibit the subject from participating in the study or may hinder the collection of data and interpretation of the results

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with primary or recurrent benign bone tumor or tumor-like condition that requires operative treatment by means of tumor evacuation and defect filling.
Sampling Method: Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2009-03 (Actual); Primary Completion 2014-02 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Stratum I: Hand-grip strength test | 3 months
  Hand and finger grip strength measured by a standard device
Stratum II: Healing of cortical bone window based on CT scan evaluation | 6 months
  CT-evaluation of cortical defect healing

SECONDARY OUTCOMES:
Biomaterial incorporation assessed with radiographs | 3, 6, and 12 months
  Radiographic evaluation of bioactive glass and bone graft incorporation
Pain intensity (VAS) | 3,6, and 12 months
  Evaluation of postoperative pain
Stratum I: DASH-questionnaire | 3,6, and 12 months
  Evaluation of patient-related outcome
RAND-36 | 3,6, and 12 months
  Evaluation of patient-related outcome
Surgical wound healing | 0-3 months
  Clinical evaluation of surgical wound healing
Soft tissue complications | 0-12 months
  Clinical evaluation of soft tissue complications in the surgical area
Bone complications | 0-12 months
  Clinical and radiographic evaluation of complications of bone defect healing

CONTACTS AND LOCATIONS:
Overall Officials: Hannu T Aro, MD, PhD, Principal Investigator — Turku University Central Hospital and University of Turku
Locations (5):
- Finland (5):
  - Helsinki University Hospital, Helsinki
  - Kuopio University Hospital, Kuopio
  - Oulu University Hospital, Oulu
  - Tampere University Hsopital, Tampere
  - Turku University Central Hospital, Turku

REFERENCES:
- [Background] Keranen P, Itala A, Koort J, Kohonen I, Dalstra M, Kommonen B, Aro HT. Bioactive glass granules as extender of autogenous bone grafting in cementless intercalary implant of the canine femur. Scand J Surg. 2007;96(3):243-51. doi: 10.1177/145749690709600310. PMID 17966751
- [Background] Valimaki VV, Aro HT. Molecular basis for action of bioactive glasses as bone graft substitute. Scand J Surg. 2006;95(2):95-102. doi: 10.1177/145749690609500204. PMID 16821652
- [Background] Valimaki VV, Moritz N, Yrjans JJ, Vuorio E, Aro HT. Effect of zoledronic acid on incorporation of a bioceramic bone graft substitute. Bone. 2006 Mar;38(3):432-43. doi: 10.1016/j.bone.2005.09.016. Epub 2005 Dec 9. PMID 16338190
- [Background] Valimaki VV, Yrjans JJ, Vuorio E, Aro HT. Combined effect of BMP-2 gene transfer and bioactive glass microspheres on enhancement of new bone formation. J Biomed Mater Res A. 2005 Dec 1;75(3):501-9. doi: 10.1002/jbm.a.30236. PMID 16116592
- [Background] Valimaki VV, Moritz N, Yrjans JJ, Dalstra M, Aro HT. Peripheral quantitative computed tomography in evaluation of bioactive glass incorporation with bone. Biomaterials. 2005 Nov;26(33):6693-703. doi: 10.1016/j.biomaterials.2005.04.033. PMID 15941582
- [Background] Koort JK, Makinen TJ, Suokas E, Veiranto M, Jalava J, Knuuti J, Tormala P, Aro HT. Efficacy of ciprofloxacin-releasing bioabsorbable osteoconductive bone defect filler for treatment of experimental osteomyelitis due to Staphylococcus aureus. Antimicrob Agents Chemother. 2005 Apr;49(4):1502-8. doi: 10.1128/AAC.49.4.1502-1508.2005. PMID 15793132
- [Background] Itala A, Koort J, Ylanen HO, Hupa M, Aro HT. Biologic significance of surface microroughing in bone incorporation of porous bioactive glass implants. J Biomed Mater Res A. 2003 Nov 1;67(2):496-503. doi: 10.1002/jbm.a.10501. PMID 14566790
- [Background] Itala A, Valimaki VV, Kiviranta R, Ylanen HO, Hupa M, Vuorio E, Aro HT. Molecular biologic comparison of new bone formation and resorption on microrough and smooth bioactive glass microspheres. J Biomed Mater Res B Appl Biomater. 2003 Apr 15;65(1):163-70. doi: 10.1002/jbm.b.10529. PMID 12632386
- [Background] Itala A, Ylanen HO, Yrjans J, Heino T, Hentunen T, Hupa M, Aro HT. Characterization of microrough bioactive glass surface: surface reactions and osteoblast responses in vitro. J Biomed Mater Res. 2002 Dec 5;62(3):404-11. doi: 10.1002/jbm.10273. PMID 12209926
- [Background] Gao T, Aro HT, Ylanen H, Vuorio E. Silica-based bioactive glasses modulate expression of bone morphogenetic protein-2 mRNA in Saos-2 osteoblasts in vitro. Biomaterials. 2001 Jun;22(12):1475-83. doi: 10.1016/s0142-9612(00)00288-x. PMID 11374446
- [Background] Itala A, Nordstrom EG, Ylanen H, Aro HT, Hupa M. Creation of microrough surface on sintered bioactive glass microspheres. J Biomed Mater Res. 2001 Aug;56(2):282-8. doi: 10.1002/1097-4636(200108)56:23.0.co;2-5. PMID 11340600
- [Background] Ylanen HO, Helminen T, Helminen A, Rantakokko J, Karlsson KH, Aro HT. Porous bioactive glass matrix in reconstruction of articular osteochondral defects. Ann Chir Gynaecol. 1999;88(3):237-45. PMID 10532567
- [Background] Virolainen P, Heikkila J, Yli-Urpo A, Vuorio E, Aro HT. Histomorphometric and molecular biologic comparison of bioactive glass granules and autogenous bone grafts in augmentation of bone defect healing. J Biomed Mater Res. 1997 Apr;35(1):9-17. doi: 10.1002/(sici)1097-4636(199704)35:13.0.co;2-s. PMID 9104694
- See also: Home site of the principal research center — http://www.orthopaedics.utu.fi